CLINICAL TRIAL: NCT05423171
Title: Predictors of Response to an Intensive Bimanual Intervention in Children With Cerebral Palsy
Brief Title: Intensive Bimanual Intervention in Cerebral Palsy Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Catherine Mercier, Full Professor, Université Laval, Scientific Director, Cirris, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Manœuvre
Record Dates: First submitted 2022-05-25; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
Keywords: Intensive bimanual therapy; Upper limb motor function; Rehabilitation; Motor learning; Accelerometry
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MANUS (Experimental): Children and youth living with cerebral palsy will take part in a 60-hour intensive bimanual therapy at Peps at Université Laval, during which they will play games and exercise to promote spontaneous use of the most affected hand. Participants will take part to pre-evaluation and 1-week and 6-month post-intervention.
  Interventions: Other: Intensive bimanual therapy

INTERVENTIONS:
Other: Intensive bimanual therapy — 60-hour intensive therapy promoting the use of both hands (ex: bimanual activities, games,...)

SUMMARY:
Motor disorders related to cerebral palsy are often accompanied by sensory, cognitive, perceptive, communication and behavioural impairments. It has already been shown that intensive bimanual intervention can improve arm movement, but its impact on the spontaneous use of the most affected arm in everyday life remains to be established. This project aims to understand the impacts of an intensive bimanual therapy on uni- and bi-manual motor functions as well as the spontaneous use of the most affected arm. Predictive value of neuroimaging variables will also be assessed.

DETAILED DESCRIPTION:
Most activities of everyday life require the use of both hands in a coordinated manner. Motor disorders related to cerebral palsy lead to activity limitations due to motor function disturbances. It has already been shown that intensive bimanual intervention can improve arm movement, but its impact on the spontaneous use of the most affected arm in everyday life remains to be established. This project aims to understand the impacts of intensive bimanual therapy on the motor functions of both arms (working together or in isolation) as well as on the spontaneous use of the most affected limb. Predictive value of neuroimaging variables will also be assessed. Thirty children living with cerebral palsy will be recruited over a 5-year period. The intervention consists of a day camp, where a small group of participants will be stimulated (one worker per child) to do activities using both hands 6 hours/day for 10 days. There will be three periods of evaluation (pre-intervention, post-intervention and 6-month follow-up). These evaluation periods consist of neuroimaging assessment, clinical evaluation, robotic evaluation and movement evaluation using inertial control units. The use of more accurate measurements of sensorimotor arm functions using robotic systems will clarify the relationship between measurements of brain function and clinical improvements, to better understand the significant variability observed in response to interventions.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of cerebral palsy or spastic hemiparesis encephalopathy
* Having sensorimotor deficits of one or both upper limb (spastic hemiparesis with a dominance on one side of the body; Manual Ability Classification System (MACS) level

  1, 2 or 3);
* Having cognitive capacities to understand and perform task of the study.

Exclusion Criteria:

* Presenting other significant health problem which may interfere with the requested task or with the clinical intervention;
* Having Botox injection in one or both upper limbs with the 4 months prior to the intervention;
* Presenting significant uncorrected visual deficits.

N.B. Having a ferromagnetic implant is not an exclusion criterion, such participant will be eligible but will not perform the MRI.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | Measured prior to the intervention.
  Neurophysiological evaluation
Robotic evaluation - Visually guided reaching | Measured prior to the intervention.
  The participant must reach as quickly and accurately as possible 4 targets spread over a radius of 10 cm around the starting target, presented in a pseudo-random order (total of 32 reaching movements)
Robotic evaluation - Visually guided reaching | Measured one week post-intervention.
  The participant must reach as quickly and accurately as possible 4 targets spread over a radius of 10 cm around the starting target, presented in a pseudo-random order (total of 32 reaching movements)
Robotic evaluation - Visually guided reaching | Measured 6-month post-intervention.
  The participant must reach as quickly and accurately as possible 4 targets spread over a radius of 10 cm around the starting target, presented in a pseudo-random order (total of 32 reaching movements)
Robotic evaluation - Object hit | Measured prior to the intervention.
  The participant must hit the balls with the hand of they choice, each successful contact generating haptic feedback.
Robotic evaluation - Object hit | Measured one week post-intervention.
  The participant must hit the balls with the hand of they choice, each successful contact generating haptic feedback.
Robotic evaluation - Object hit | Measured 6-month post-intervention.
  The participant must hit the balls with the hand of they choice, each successful contact generating haptic feedback.
Robotic evaluation - Ball on bar | Measured prior to the intervention.
  Four targets are successively presented to the participant, the objective of the task is to move the ball into each target as quickly and accurately as possible.
Robotic evaluation - Ball on bar | Measured one week post-intervention.
  Four targets are successively presented to the participant, the objective of the task is to move the ball into each target as quickly and accurately as possible.
Robotic evaluation - Ball on bar | Measured 6-month post-intervention.
  Four targets are successively presented to the participant, the objective of the task is to move the ball into each target as quickly and accurately as possible.
Robotic evaluation - Arm-position matching | Measured prior to the intervention.
  In this proprioception task the sense of upper limb position is evaluated
Robotic evaluation - Arm-position matching | Measured one week post-intervention.
  In this proprioception task the sense of upper limb position is evaluated
Robotic evaluation - Arm-position matching | Measured 6-month post-intervention.
  In this proprioception task the sense of upper limb position is evaluated
Spontaneous use of both arms | Measured during two-days prior to the intervention.
  The unilateral and bilateral functions will be quantified by summing the activities detected at the upper limbs with accelerometers, allowing to obtain use-ratio of each limb.
Spontaneous use of both arms | Measured two days during the intervention.
  The unilateral and bilateral functions will be quantified by summing the activities detected at the upper limbs with accelerometers, allowing to obtain use-ratio of each limb.
Spontaneous use of both arms | Measured during two-days one week post-intervention.
  The unilateral and bilateral functions will be quantified by summing the activities detected at the upper limbs with accelerometers, allowing to obtain use-ratio of each limb.
Spontaneous use of both arms | Measured during two-days 6-month post-intervention.
  The unilateral and bilateral functions will be quantified by summing the activities detected at the upper limbs with accelerometers, allowing to obtain use-ratio of each limb.
Clinical evaluation -Two-point discrimination test (TPDT) | Measured prior to the intervention.
  Sensitive test to determine tactile threshold
Clinical evaluation -Two-point discrimination test (TPDT) | Measured one week post-intervention.
  Sensitive test to determine tactile threshold
Clinical evaluation -Two-point discrimination test (TPDT) | Measured 6-month post-intervention.
  Sensitive test to determine tactile threshold.
Clinical evaluation - Jebsen Taylor Test of Hand Function (JTTHF) | Measured prior to the intervention.
  Seven standardized tasks to evaluate the unimanual function. 6 tasks. Sub-task score is the time to complete the task (a maximum of 120s is allowed per task) and the total score is the total time to perform the six tasks (maximum of 720s). Higher time means worse outcome.
Clinical evaluation - Jebsen Taylor Test of Hand Function (JTTHF) | Measured one week post-intervention.
  Seven standardized tasks to evaluate the unimanual function. 6 tasks. Sub-task score is the time to complete the task (a maximum of 120s is allowed per task) and the total score is the total time to perform the six tasks (maximum of 720s). Higher time means worse outcome.
Clinical evaluation - Jebsen Taylor Test of Hand Function (JTTHF) | Measured 6-month post-intervention.
  Seven standardized tasks to evaluate the unimanual function
Clinical evaluation - Box and Blocks Test (BBT) | Measured prior to the intervention.
  Measurement of manual dexterity of each hand. The participant must take one block at a time with one hand to transfer it to the other side of the box.
Clinical evaluation - Box and Blocks Test (BBT) | Measured one week post-intervention.
  Measurement of manual dexterity of each hand. The participant must take one block at a time with one hand to transfer it to the other side of the box.
Clinical evaluation - Box and Blocks Test (BBT) | Measured 6-month post-intervention.
  Measurement of manual dexterity of each hand. The participant must take one block at a time with one hand to transfer it to the other side of the box.
Clinical evaluation - Assisting Hand Assessment (AHA) | Measured prior to the intervention.
  This test consists of standardized tasks with toys during a semi-structured game session. The test is recorded, and the video is analyzed and scored later. Logit-based 0 to 100 AHA-unit scale (score 0-100; better score means better outcome).
Clinical evaluation - Assisting Hand Assessment (AHA) | Measured one week post-intervention.
  This test consists of standardized tasks with toys during a semi-structured game session. The test is recorded, and the video is analyzed and scored later. Logit-based 0 to 100 AHA-unit scale (score 0-100; better score means better outcome).
Clinical evaluation - Assisting Hand Assessment (AHA) | Measured 6-month post-intervention.
  This test consists of standardized tasks with toys during a semi-structured game session. The test is recorded, and the video is analyzed and scored later. Logit-based 0 to 100 AHA-unit scale (score 0-100; better score means better outcome).
Clinical evaluation - Two-Arm Coordination Test (TACT) | Measured prior to the intervention.
  Evaluation of the constrained bilateral use of both upper limbs with an electronic tracking device (eight tests; four clockwise and four counter-clockwise).
Clinical evaluation - Two-Arm Coordination Test (TACT) | Measured one week post-intervention.
  Evaluation of the constrained bilateral use of both upper limbs with an electronic tracking device (eight tests; four clockwise and four counter-clockwise).
Clinical evaluation - Two-Arm Coordination Test (TACT) | Measured 6-month post-intervention.
  Evaluation of the constrained bilateral use of both upper limbs with an electronic tracking device (eight tests; four clockwise and four counter-clockwise).
Clinical evaluation - Motor-Free Visual Perception Test-Revised (MVPT-R) | Measured prior to the intervention.
  Visual perception test that assesses consistency of form, spatial orientation, discrimination, memory and visual closure (Score: 0 - 40; better score means better outcome).
Clinical evaluation - Motor-Free Visual Perception Test-Revised (MVPT-R) | Measured one week post-intervention.
  Visual perception test that assesses consistency of form, spatial orientation, discrimination, memory and visual closure (Score: 0 - 40; better score means better outcome).
Clinical evaluation - Motor-Free Visual Perception Test-Revised (MVPT-R) | Measured 6-month post-intervention.
  Visual perception test that assesses consistency of form, spatial orientation, discrimination, memory and visual closure (Score: 0 - 40; better score means better outcome).

SECONDARY OUTCOMES:
Self-assessments - Children's Hand-use Experience Questionnaire (CHEQ) | Measured prior to the intervention.
  CHEQ is a 29 item child-completed questionnaire that examines how the weaker/affected limb is used in everyday activities. It presents a list of common daily activities that typically require use of two hands. The child then rates the time required, the efficacy of grasp, and how bothered they feel by their hand function on the task. Total score transformed by a Rasch analysis into a scale of 0-100 units (better score means better outcome).
Self-assessments - Children's Hand-use Experience Questionnaire (CHEQ) | Measured one week post-intervention.
  CHEQ is a 29 item child-completed questionnaire that examines how the weaker/affected limb is used in everyday activities. It presents a list of common daily activities that typically require use of two hands. The child then rates the time required, the efficacy of grasp, and how bothered they feel by their hand function on the task. Total score transformed by a Rasch analysis into a scale of 0-100 units (better score means better outcome).
Self-assessments - Children's Hand-use Experience Questionnaire (CHEQ) | Measured 6-month post-intervention.
  CHEQ is a 29 item child-completed questionnaire that examines how the weaker/affected limb is used in everyday activities. It presents a list of common daily activities that typically require use of two hands. The child then rates the time required, the efficacy of grasp, and how bothered they feel by their hand function on the task. Total score transformed by a Rasch analysis into a scale of 0-100 units (better score means better outcome).
Self-assessments - Canadian Occupational Performance Measure (COPM) | Measured prior to the intervention.
  Prior to the intervention, children, parents and therapists will work together to set a therapy goal related to their hand or wrist function. The child will score their current performance/satisfaction on the identified activity and will re-score post-intervention. Performance: scale from 0 to 10, better the score is better is the outcome. Satisfaction: scale from 0 to 10, better the score is better is the outcome.
Self-assessments - Canadian Occupational Performance Measure (COPM) | Measured one week post-intervention.
  Prior to the intervention, children, parents and therapists will work together to set a therapy goal related to their hand or wrist function. The child will score their current performance/satisfaction on the identified activity and will re-score post-intervention.Performance: scale from 0 to 10, better the score is better is the outcome. Satisfaction: scale from 0 to 10, better the score is better is the outcome.
Self-assessments - Canadian Occupational Performance Measure (COPM) | Measured 6-month post-intervention.
  Prior to the intervention, children, parents and therapists will work together to set a therapy goal related to their hand or wrist function. The child will score their current performance/satisfaction on the identified activity and will re-score post-intervention. Performance: scale from 0 to 10, better the score is better is the outcome. Satisfaction: scale from 0 to 10, better the score is better is the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Université Laval, Québec, Canada

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT05423171/Prot_SAP_000.pdf
  • Informed Consent Form: First participation (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT05423171/ICF_001.pdf
  • Informed Consent Form: Second participation and more (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT05423171/ICF_002.pdf